CLINICAL TRIAL: NCT05533788
Title: A Randomized, Open-label, Two Sequence, Two-period Cross-over Study Evaluating the Relative Bioavailability of ABSK091 Single Dose Between Fed and Fasted States in Healthy Subjects
Brief Title: ABSK091 Food Effect Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: ABSK091-101
Record Dates: First submitted 2021-10-11; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Health, Subjective; Food-drug Interaction
MeSH Terms: interventions — AZD4547

STUDY DESIGN:
Intervention Model Description: In this study, a single oral dose of the tablet formulation administered under fed conditions will be compared to administration under fasted conditions to assess the effects of high-fat meal on the rate and extent of absorption and exposure.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fed states in healthy subjects (Other): Fed states in healthy subjects
  Interventions: Drug: ABSK091 tablet
- Fasted states in healthy subjects (Other): Fasted states in healthy subjects
  Interventions: Drug: ABSK091 tablet

INTERVENTIONS:
Drug: ABSK091 tablet — ABSK091 tablet which is being developed for the treatment of patients with advanced solid tumors
  Other Names: AZD4547 tablet

SUMMARY:
In this study, a single oral dose of the tablet formulation administered under fed conditions will be compared to administration under fasted conditions to assess the effects of a high-fat meal on the rate and extent of absorption and exposure.

Study ABSK091-101 is a single-center, Phase 1, open-label, randomized, two-period, two-sequence, and crossover study in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent prior to any study specific procedures
2. aged 20 to 45 years, inclusive, at the time of screening
3. male subjects: agree to use an effective method of contraception and not donate sperm for the duration of the study and for 3 months following the last dose of ABSK091
4. female subjects: non-pregnant, non-lactating female subjects who if premenopausal are using adequate birth control, e.g., oral, injectable, transdermal or implanted hormonal contraceptives, vaginal contraceptive ring, intrauterine device/intrauterine system, tubal ligation, vasectomized sexual partner (with confirmed negative sperm counts) or true sexual abstinence. All females must have a negative serum pregnancy test within 7 days and a negative urine pregnancy test within 24 hours prior to dosing with ABSK091
5. have a body mass index (BMI) of 18.5 to 24.9 kg/m2, inclusive, and weigh at least 50 kg and no more than 90 kg, at screening
6. healthy subjects as determined by medical history and physical examination and have clinical laboratory test results within normal reference range for the investigative site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
7. with suitable veins for cannulation or repeated vein puncture
8. are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

1. Are currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
2. Have participated, within the last 30 days, in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed.
3. Have previously completed or withdrawn from this study or any other study investigating ABSK091, and have previously received the investigational product
4. Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
5. Have known allergies to ABSK091, related compounds, or any components of the formulation, or history of significant atopy.
6. Have known or ongoing psychiatric disorders that would interfere with study participation as determined by the investigator.
7. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of ABSK091 .
8. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results as judged by the Investigator.
9. Have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participating in the study.
10. Prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 ms (female >480 ms) or shortened QTcF <350 ms or family history of long QT syndrome.
11. Have an abnormal blood pressure as determined by the investigator.
12. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody and human immunodeficiency virus (HIV) .
13. Any of the following ophthalmological criteria.
14. Known or suspected history of drug abuse as judged by the Investigator.
15. Have used or intend to use over-the-counter or prescription medication , including herbal medications, within 14 days prior to dosing and during the study
16. Plasma donation within one month of screening or any blood. donation/blood loss >500 mL during the 3 months prior to screening
17. Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or are unwilling to abide by alcohol restrictions as specified in Section 6.3.2 (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
18. are subjects who currently smoke more than 5 cigarettes per day (or equivalent in tobacco or nicotine products) or are unwilling to abide by smoking restrictions as specified in Section 6.3.2
19. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade or other products containing grapefruit or Seville oranges within 7 days before the first administration of the ABSK091
20. have a current or recent history (<30 days prior to screening and/or <45 days prior to Day -1 in Period 1) of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection
21. have had symptomatic herpes zoster within 3 months of screening
22. have received live vaccine(s) within 3 months of screening, or intend to during the study
23. are unwilling to comply with the dietary requirements/restrictions during the study.
24. have used or intend to use drugs or substances that are known to be strong or moderate inhibitors or inducers of CYP 3A4/5 and/or CYP2D6 within 30 days prior to the first dose and throughout the study.
25. Have a history of, in the opinion of the investigator, excessive methylxanthine use within the previous 6 months, or are unwilling to abide by restrictions as specified in Section 6.3.2. Excessive intake is defined as more than 6 units of caffeine per day; one caffeine unit is contained in the following items: 1 (177 mL) cup of coffee, 1 (355 mL) cup of tea, 2 (355 mL) cans of cola, or 3 oz (85 g) of chocolate
26. Involvement in the planning and/or conduct of the study (applies to Abbisko staff, CRO staff, and staff at the study site)
27. in the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Cmax | 9 days
  The PK parameters of Cmax
AUC(0-tlast) | 9 days
  The PK parameters of AUC(0-tlast)
AUC(0-∞) | 9 days
  The PK parameters of AUC(0-∞)
Tmax | 9 days
  The PK parameters of Tmax

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | 9 days
  Incidence and severity of treatment-emergent adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Lu, PhD, Study Director — Abbisko Therapeutics Co, Ltd
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided